CLINICAL TRIAL: NCT03469141
Title: Interactive Telehealth and Auto-Biofeedback Sensor System for Pressure Ulcer Prevention After SCI
Brief Title: Interactive Telehealth for Pressure Ulcer Prevention After SCI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rancho Research Institute, Inc. (Other)
Responsible Party: Principal Investigator, Sara Mulroy, Co-Director, Rancho Research Institute, Inc.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 90SI5018
Record Dates: First submitted 2018-03-12; First posted 2018-03-19 (Actual); Last update posted 2018-06-13 (Actual); Status verified 2018-06

CONDITIONS: Spinal Cord Injuries; Pressure Ulcer
Keywords: Wheelchair; Pressure Relief; Activity; Monitor
MeSH Terms: conditions — Spinal Cord Injuries; Pressure Ulcer; Motor Activity

STUDY DESIGN:
Intervention Model Description: All participants will complete two weeks of recording PR behavior by the monitoring system without feedback. Following baseline assessment, participants will be randomized into one of two groups: an intervention group that will receive an education session on PU prevention with goal setting for PR frequency and duration followed by four weeks of biofeedback via the smartphone app component of the monitoring system, or a control group that will receive only the education and goal setting session, but will not receive biofeedback and will have the WC sensor system for measurement only. After four weeks, the biofeedback feature in the intervention group will be turned off. The system will continue to monitor activities for another two weeks. We will assess whether improvements in PR adherence are retained after the 4-week bout of biofeedback (washout). Participants will return one year following the 8-week intervention to assess whether they have developed a PU.
Who Masked: Participant
Masking Description: Following the training/goal setting session, participants will be randomly assigned into either the intervention group that will receive biofeedback via the smartphone app for 4 weeks, or the control group that will continue to have the WC sensor system for measurement only and will not receive biofeedback.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Control Group (No Intervention): The control group will continue to have the WC sensor system for measurement only and will not receive biofeedback after receiving instructions on the importance of pressure relief (PR) maneuvers for skin care, as well as training regarding the three pressure relief maneuvers. Materials (including fact sheets, etc.) will be incorporated in the educational content of the project.
- Intervention Group (Experimental): The intervention group will receive biofeedback via the smartphone app.
  Interventions: Device: Pressure Relief Monitoring System

INTERVENTIONS:
Device: Pressure Relief Monitoring System — Biofeedback provided to the intervention group via the smartphone app will include: Visual (e.g., phone notification bar) and auditory reminders if PR (pressure relief) is not performed as scheduled, Real-time feedback during performance of PR maneuvers to ensure adequate PR (e.g., the app will indicate if the duration of PR is sufficient), and Aggregate counts of daily PR activity.
  Other Names: Sensimat
  Arms: Intervention Group

SUMMARY:
The goal of this module project is to establish the efficacy of a portable sensor and app-based biofeedback technology system for promoting effective pressure relief behaviors and reducing risk of pressure ulcer development among wheelchair users. In collaboration with the participating SCIMS centers, the investigators will conduct a randomized clinical trial of education and goal setting alone compared to education and goal setting combined with the biofeedback system (SENSIMAT®) that is commercially available.

DETAILED DESCRIPTION:
Overview and Rationale:

Pressure ulcers (PUs) are a frequent and serious secondary complication after SCI with an annual incidence of 31% and a lifetime incidence of up to 85%. PUs are linked to increased morbidity and mortality. As medical or surgical repair of established PUs is difficult and costly, the preferred approach is prevention. Traditional prevention recommendations included intermittent relief of interface pressure, such as performing wheelchair (WC) pushups every 30 minutes for 30 seconds or once an hour for 60 seconds. Alternatives to the push-up maneuver, including forward and lateral trunk leans, have been recommended to reduce the demands of weight bearing on the shoulders. One approach to address inadequate PR is to provide a simple reminder (i.e., an alarm) at set intervals. However, this approach is inadequate because patients who attempt PR maneuvers often do not achieve an adequate magnitude or duration of PR for tissue unloading. In addition, compliance with PR performance can be negatively impacted by unanticipated life circumstances. A system to measure PR maneuvers in the home and community and provide reminders and feedback on frequency and success of individual attempts of this important preventative activity could reduce the incidence of PUs. In this collaborative project, the investigators will establish the efficacy of a sensor and feedback technology system for promoting effective pressure relief behaviors and reducing risk of pressure ulcer development among wheelchair users. The investigators will conduct a randomized clinical trial of education and goal setting alone compared to education and goal setting combined with the biofeedback system (sensor and smartphone app) that is developed and validated. The fully functional system is unobtrusive and simple. The system attaches to any WC (without modification) and generates automatic reminders via an app. Biofeedback, also delivered via the app, indicates in real time when a PR maneuver has been completed successfully. The display also tracks the user's daily PR activity as the participants works towards a daily goal.

Specific Aims:

Primary: Compare PR behavior (daily PR frequency and average duration of uninterrupted sitting) between participants who receive education and four weeks of biofeedback training with the monitoring system (intervention group) and those who receive education but no system feedback (control group). Secondary: Compare the incidence of ischial PU development at one year post-intervention between groups.

Hypotheses:

1) Biofeedback from the monitoring system will increase PR frequency and decrease uninterrupted sitting time compared to that achieved by education and goal setting without feedback. 2) Improvements in PR adherence will be retained after two weeks of wash-out (no feedback). 1) Incidence of ischial PU development will be lower in participants who receive feedback training with the telehealth monitoring system than in the control group. Methods: Participants will be at least 18 years of age, between 2 and 6 months post SCI, full-time WC users for community mobility (AIS A-C), able to perform PR maneuvers without assistance, and have no current or prior history of a PU. A total of one hundred (n=100) manual WC users from all collaborating centers will participate in an 8-week monitoring trial with a one-year follow-up to assess PU development. All participants will complete two weeks of recording PR behavior by the monitoring system without feedback. Following baseline assessment, participants will be randomized into one of two groups: an intervention group that will receive an education session on PU prevention with goal setting for PR frequency and duration followed by four weeks of biofeedback via the smartphone app component of the monitoring system, or a control group that will receive only the education and goal setting session, but will not receive biofeedback and will have the WC sensor system for measurement only. After four weeks, the biofeedback feature in the intervention group will be turned off. The system will continue to monitor activities for another two weeks. The investigators will assess whether improvements in PR adherence are retained after the 4-week bout of biofeedback (washout). Participants will return one year following the 8-week intervention to assess whether they have developed a PU. Participants will be queried and their medical record reviewed regarding PU occurrence since the intervention. A physician, nurse, or other clinician will examine participants' skin visually and record presence of any PUs (stages 1-4) in the ischial region.

Proposed Outcomes:

To establish the efficacy of the wheelchair seat sensor and app-based biofeedback for establishing healthy self-management behaviors (pressure relief maneuvers) and reducing incidence of pressure ulcer development in individuals with recent SCI.

ELIGIBILITY:
Inclusion Criteria:

* Persons with documented SCI, American Spinal Injury Association Impairment Scale (AIS) A, B, or C.
* Persons who are full time manual wheelchair users.
* persons over the age of 18.
* 2-6 months post-injury.
* Able to perform pressure relief maneuvers without assistance
* Cognitively able to understand and sign informed consent form approved by the IRB
* Free of shoulder pain that interferes with daily activities or requires medical intervention at the time of enrollment in the study

Exclusion Criteria:

* History of shoulder injury or surgery or orthopedic or neurologic disorders (other than SCI) that would impact arm function, preventing them from performing pressure ulcer relief maneuvers or propelling a wheelchair.
* history of ischial pressure ulcer.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2020-10-30 (Estimated); Study Completion 2021-10-30 (Estimated)

PRIMARY OUTCOMES:
PR maneuvers per day | 8 weeks
  Number of pressure relief maneuvers per day
Sitting time | 8 weeks
  Duration of uninterrupted sitting time in minutes per day

SECONDARY OUTCOMES:
Pressure Ulcer Occurence | 1 year
  Incidence of ischial pressure ulcer occurence after one year

CONTACTS AND LOCATIONS:
Overall Officials: Sara J Mulroy, PhD,PT, Study Director — Rancho Los Amigos National Rehabilitation Center
Locations (4):
- United States (4):
  - University of Alabama, Birmingham, Alabama
  - Rancho Los Amigos National Rehabilitation Center, Downey, California
  - University of Miami, Miami, Florida
  - Thomas Jefferson University, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided
De-identified primary and secondary outcomes data will be shared with collaborators